CLINICAL TRIAL: NCT05819034
Title: Orthotic Management for Controlling Scoliotic Curve Progression in Adolescent Idiopathic Scoliosis
Brief Title: Conservative Management for Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSR02
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis; Adolescence
Keywords: Adolescents Idiopathic Scoliosis; Physical Therapy; Orthosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Adolescents in the control group will receive a scoliosis-specific exercise program which will be prescribed to control the progression of the scoliotic curve
  Interventions: Other: Scoliosis-Specific Exercise Program
- Experimental Group (Experimental): Adolescents in the experimental group will receive a scoliosis-specific exercise program which will be prescribed to control the progression of the scoliotic curve in addition to wearing the soft orthoses with external strapping.
  Interventions: Other: Scoliosis-Specific Exercise Program; Other: Soft orthoses with external strapping.

INTERVENTIONS:
Other: Scoliosis-Specific Exercise Program — Adolescents in the control group will receive a scoliosis-specific exercise program which will be prescribed to control the progression of the scoliotic curve. This exercise program will include frontal plane active or passive correction exercises for scoliotic posture. The exercise program for every participant will be three sessions per week for 12 successive weeks. Every treatment session was applied for one hour.The exercise program for every participant will be three sessions per week for 12 successive weeks. Every treatment session was applied for one hour.
  The exercise program for every participant will be three sessions per week for 12 successive weeks. Every treatment session was applied for one hour.
Other: Soft orthoses with external strapping. — Adolescents in the experimental group will receive a scoliosis-specific exercises program which will be prescribed to control the progression of the scoliotic curve in addition to wearing the soft orthoses with external strapping. The wearing schedule of the soft orthosis with the external strapping for every participant in this group will be 12 hours daily for 12 successive weeks.
  Arms: Experimental Group

SUMMARY:
Idiopathic scoliosis is a living problem that resists correction. The underlying cause of the such disorder is unknown but directed more toward muscular disorders. However recent clinical observation showed a possible neuromuscular compromise early in those patients. The main purpose of this study is to develop a treatment procedure to correct the degree of bony curvature in patients with Idiopathic scoliosis through developing a neuromuscular corrective approach that might be a more effective conservative treatment protocol for such disorder.

DETAILED DESCRIPTION:
Scoliosis is one of the most common spinal deformities occurring in school-going children during the growth spurts of adolescents. It is an abnormal curvature of the spine. Failure of early management of idiopathic scoliosis could lead to multiple problems related to postural malalignment, pulmonary and physical dysfunctions, and surgical interventions. These problems could lead to health-related quality-of-life issues such as psychological and social problems that are represented in social isolation, depression, loss of self-confidence, limited job opportunities, and hospital stays & days off school and university as a result of undergoing corrective surgeries. Treatment methods for adolescent idiopathic Scoliosis (AIS) vary between surgical intervention and conservative treatment, in mild and moderate cases. Conservative treatment includes physical therapy in addition to rigid splints and braces, which may cause pain, tightness, restriction of movement, and a bad psychological status for adolescents which may lead them to the irregular wearing of these splints and braces. A type of soft, lightweight, breathable orthosis which is TheraTogs orthotic undergarment with the strapping system has been fabricated to provide gentle, passive compression to correct spinal deformities. Therefore, the objective of this study is to evaluate the effectiveness of TheraTogs orthotic undergarment with the strapping system on controlling and modulating the degree of scoliosis in Saudi adolescents with idiopathic scoliosis.

ELIGIBILITY:
The inclusion criteria will be:

* Adolescents of both sexes with an age range between 10-17 years.
* They were diagnosed with Adolescent idiopathic scoliosis by an orthopedic specialist, confirmed through (loaded) X- rays.
* They have mild non-structural scoliosis with Cobb's angle measurement of between 10 and 25 degrees
* They have Single major thoracolumbar curve located between T6-7 to L1-2, apex at T12 or L1.
* They have good health conditions except for scoliosis.
* They can understand and communicate with no mental abnormalities.

The exclusion criteria will be:

* Adolescents with cerebral palsy or other degenerative neurological disorders;
* Participants with nutritional disorders e.g. diabetes or vascular disorders.
* Participants with a scoliotic curve with angle > 25° will be excluded.
* Participants will be excluded from this study if they have inflexible spinal deformities interfering with spinal mobility,
* Participants who were subjected to any corrective surgery to their spine within the previous two years.
* Participants will be also excluded if their skin were sensitive or inflamed to any materials used.
* Participants who have seizures, perceptual disorders, visual problems, and auditory deficits
* Participants who have leg length discrepancy
* Participants who have scoliosis developed as a consequence of traumatic scoliosis.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in the scoliotic cobb's angle (°) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  X-ray imaging will be measured by a radiologist
Changes in the Pelvic Obliquity (mm) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The following device (DIERS Formetric 3D/4D spine & posture analysis system) will be used to examine the changes in the spinal vertebral parameters in different planes (sagittal, coronal and transverse). This device supplies a thorough report about the alignment of the whole spine in one assessment session.
Change in the vertebral rotation (Angle) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The following device (DIERS Formetric 3D/4D spine & posture analysis system) will be used to examine the changes in the spinal vertebral parameters in different planes (sagittal, coronal and transverse). This device supplies a thorough report about the alignment of the whole spine in one assessment session.
Change in the Coronal imbalance (mm) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The following device (DIERS Formetric 3D/4D spine & posture analysis system) will be used to examine the changes in the spinal vertebral parameters in different planes (sagittal, coronal and transverse). This device supplies a thorough report about the alignment of the whole spine in one assessment session.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab M Abd El Kafy, PhD, Principal Investigator — Department of Physical Therapy- Faculty of Applied Medical Sciences - Umm Al Qura University
Locations (1):
- Umm Al Qura University, Mecca, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
- The data available is Case-by-case basis at the discretion of the Primary Sponsor
Supporting Information: SAP
Time Frame: Start Date: Beginning one year following main results publication End Date: Ending two years following main results publication
Access Criteria: Data can be obtained by Principal Investigator Email Address: emkafy@uqu.edu.sa